CLINICAL TRIAL: NCT04848220
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Effect on Microvascular Obstruction of Temanogrel in Subjects Undergoing Percutaneous Coronary Intervention
Brief Title: A Study Evaluating the Safety, Tolerability, and Effect on Microvascular Obstruction of Intravenous Temanogrel in Adult Participants Undergoing Percutaneous Coronary Intervention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD791-202; C5071002 (Other: Alias Study Number)
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Microvascular Obstruction
Keywords: Temanogrel; Microvascular obstruction; APD791; Percutaneous coronary intervention; MVO; PCI
MeSH Terms: interventions — APD791

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stage A (Dose Cohort 1) and Stage B (Dose Group 1) (Experimental)
  Interventions: Drug: Temanogrel
- Stage A (Dose Cohort 2) and Stage B (Dose Group 2) (Experimental)
  Interventions: Drug: Temanogrel
- Stage A (Dose Cohort 1 and Dose Cohort 2) and Stage B (Dose Group 1 and Dose Group 2) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Temanogrel — Participants will receive a single intravenous dose of temanogrel on Day 1 (Day 1 of PCI procedure)
  Arms: Stage A (Dose Cohort 1) and Stage B (Dose Group 1); Stage A (Dose Cohort 2) and Stage B (Dose Group 2)
Drug: Placebo — Participants will receive a single intravenous dose of temanogrel matching placebo on Day 1
  Arms: Stage A (Dose Cohort 1 and Dose Cohort 2) and Stage B (Dose Group 1 and Dose Group 2)

SUMMARY:
The purpose of this study is to determine whether intravenous temanogrel is a safe and effective treatment for microvascular obstruction (MVO) in adult participants undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to be conducted in 2 stages (Stage A and Stage B). Stage A is an ascending single-dose placebo-controlled study planned to consist of 2 cohorts. Stage B is a parallel-treatment group study planned to consist of a placebo group and 2 active treatment groups of temanogrel doses selected based on safety and tolerability data in Stage A.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina participants suitable for elective PCI, or participants suitable for PCI for diagnosis of non-ST-elevation myocardial infarction or unstable angina (NSTEMI/UA) who are consistently hemodynamically stable until the time of PCI and have a thrombolysis in myocardial infarction (TIMI) Flow Grade 2 or 3 on the diagnostic angiography
* Target lesions for PCI must appear suitable for stenting as confirmed on the diagnostic angiography and must satisfy the study criteria regarding lesion size and vessel diameter/type.
* Females must not be of childbearing potential
* Males with pregnant or non-pregnant female partners of childbearing potential must agree to using a condom during treatment and for 90 days following treatment

Exclusion Criteria:

* Planned or anticipated use of rotational atherectomy/ablation or shockwave therapies during the PCI procedure
* Any history of stroke, seizure, intracranial bleeding, or intracranial aneurysm
* Transient ischemic attack within the 6 months prior to Screening
* History of major trauma, major surgery, and/or clinically significant head injury or hemorrhage within the last 6 months of Screening
* Any ST-elevation myocardial infarction (STEMI) within 10 days of Screening or STEMI within the target vessel territory within the last 4 months of Screening

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (3):
  - Tibor Rubin VA Medical Center, Long Beach, California
  - VA Palo Alto - Cardiac Catheterization Laboratory, Palo Alto, California
  - University of Chicago Medical Center, Chicago, Illinois
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Alfred Health - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maasstad Hospital, Rotterdam, South Holland
  - Catharina Ziekenhuis, Eindhoven
- Skåne University Hospital, Lund, Sweden
- East and North Hertfordshire NHS Trust Lister Hospital, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD791-202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in two stages: Stage A (an ascending single dose study consisting of 2 cohorts of 20 and 40 milligram [mg] doses of temanogrel or placebo) and Stage B: parallel group study (consisting of 3 treatment groups of temanogrel 20 mg, temanogrel 40 mg and placebo). The study was terminated early due to business decision. Analysis of stage A and B was combined as pre specified in the protocol.
Pre-assignment Details: A total of 29 participants were enrolled and randomized in the study.
Groups:
- Temanogrel 20 mg: Participants received a single intravenous (IV) dose of temanogrel 20 mg on Day 1 following which the participants underwent percutaneous coronary intervention (PCI). Participants had a follow-up phone call 7 days after administration of study treatment.
- Temanogrel 40 mg: Participants received a single IV dose of temanogrel 40mg on Day 1 following which the participants underwent PCI. Participants had a follow-up phone call 7 days after administration of study treatment.
- Placebo: Participants received a single IV dose of placebo on Day 1 following which the participants underwent PCI. Participants had a follow-up phone call 7 days after administration of study treatment.
Period: Overall Study
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Started | 10 | 10 | 9
Treated | 10 | 8 | 9
Completed | 10 | 8 | 9
Not Completed | 0 | 2 | 0
Not completed — Unable to proceed to study procedure | 0 | 1 | 0
Not completed — Fractional flow not significant | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants, irrespective of whether they received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (7.81) | 64.5 (3.27) | 63.3 (9.63) | 64.6 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 9 | 10 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 8 | 9 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Index of Microcirculatory Resistance (IMR) From Baseline to Post Percutaneous Coronary Intervention (PCI)
Description: IMR was defined as the mean distal pressure at maximum hyperemia multiplied by the mean hyperemic transit time. IMRcorr (IMR corrected for the influence from collateral supply) was calculated using the following equation, to account for the presence of significant epicardial stenosis without the need for balloon dilation to measure the coronary wedge pressure (Pw), IMRcorr = mean aortic pressure at maximum hyperemia (Pa)*mean transit time at maximal hyperemia (Tmn) * [1.34 * mean distal coronary pressure at maximum hyperemia (Pd)/Pa minus 0.32].
Time Frame: From Baseline (prior to administration of study treatment) to 15 minutes post-PCI on Day 1
Population: FAS included all randomized participants, irrespective of whether they received any study treatment. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury*seconds
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9
Millimeter of mercury*seconds | -8.1783 (15.35531) | 0.0691 (13.27702) | -1.8907 (18.82659)

2. Secondary Outcome: Change From Baseline to Post-PCI for Coronary Flow Reserve (CFR)
Description: The coronary flow reserve (CFR) was calculated from the ratio of baseline (i.e., resting transit time) to hyperemic mean transit time.
Time Frame: From Baseline (prior to administration of study treatment) to 15 minutes post-PCI on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9
Ratio | 1.2744 (0.89307) | 1.0238 (2.97729) | 1.3787 (1.40440)

3. Secondary Outcome: Change From Baseline to Post-PCI for Fractional Flow Reserve (FFR)
Description: The FFR was calculated from the ratio of distal to proximal mean pressures at maximal hyperemia (FFR = [distal coronary pressure/aortic pressure at maximum hyperemia]).
Time Frame: From Baseline (prior to administration of study treatment) to 15 minutes post-PCI on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9
Ratio | 0.1346 (0.19620) | 0.2494 (0.20758) | 0.3123 (0.16562)

4. Secondary Outcome: Change From Baseline to Post-PCI for Corrected Thrombolysis in Myocardial Infarction Frame Count (cTFC)
Description: The cTFC is a quantitative index of coronary flow and was calculated based upon the number of cine-frames that the intracoronary dye required to reach distal coronary landmarks.
Time Frame: From Baseline (prior to administration of study treatment) to 15 minutes post-PCI on Day 1
Population: Safety set included all participants in the FAS who received any study treatment. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Frames per second
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 9 | 7 | 8
Frames per second | -6.54 (7.365) | -0.81 (6.320) | -8.93 (8.368)

5. Secondary Outcome: Number of Participants According to Change From Baseline to Post-PCI for Thrombolysis in Myocardial Infarction (TIMI) Flow Grade (TFG) Post-PCI
Description: The TFG is a measure of epicardial perfusion and was graded on a standard scale from 0 to 3, where Grade 0=no perfusion, grade 1=penetration without perfusion, grade 2=partial perfusion and grade 3= complete perfusion.
Time Frame: Baseline (prior to administration of study treatment) and anytime between 0 to 15 minutes post-PCI on Day 1
Population: Safety set included all participants in the FAS who received any study treatment. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  Baseline Grade 3 | 10 | 8 | 9
  0 to 15 min post-PCI Grade 3 | 9 | 8 | 8
  0 to 15 min post-PCI missing | 1 | 0 | 1

6. Secondary Outcome: Number of Participants According to Change From Baseline to Post-PCI in Thrombolysis in Myocardial Infarction Myocardial Perfusion Grade (TMPG) Post-PCI
Description: The TMPG (also known as myocardial blush grade [MBG]), is a measure of myocardial perfusion in the capillary bed at the tissues level following contrast injection into the coronary artery. TMPG was graded on a scale from 0 to 3, where grade 0 = failure of dye to enter the microvasculature; grade 1 = dye slowly enters but fails to exit the microvasculature; grade 2 = delayed entry and exit of dye from the microvasculature; grade 3= normal entry and exit of dye from the microvasculature.
Time Frame: Baseline (prior to administration of study treatment) and anytime between 0 to 15 minutes post-PCI on Day 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  Baseline TMPG value 2 | 1 | 0 | 1
  Baseline TMPG value 3 | 7 | 4 | 3
  Baseline Missing | 2 | 4 | 5
  0 to 15 min post-PCI TMPG value 3 | 9 | 6 | 6
  0 to 15 min post-PCI Missing | 1 | 2 | 3

7. Secondary Outcome: Change From Baseline to Post-PCI for Creatine Kinase (CK)
Time Frame: Baseline (prior to administration of study treatment), anytime between 0 to 15 minutes, 6 hours post-PCI, and 24 hours post-PCI/discharge
Population: Safety Set included all participants in the FAS who received any study treatment. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoints. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Units per liter
  0 to 15 minutes post-PCI | -11.7 (11.25) | -6.0 (5.68) | -5.9 (10.58)
  6 hours post-PCI: number analyzed (Participants) | 9 | 8 | 6
  6 hours post-PCI | 0.9 (17.20) | 1.5 (27.07) | -23.5 (41.03)
  24 hours post- PCI/discharge: number analyzed (Participants) | 6 | 1 | 3
  24 hours post- PCI/discharge | -33.7 (23.42) | 233.0 (NA) — Standard deviation could not be calculated for only one participant. | -6.0 (38.94)

8. Secondary Outcome: Change From Baseline to Post-PCI for Creatine Kinase-Myocardial Band (CK-MB)
Time Frame: Baseline (prior to administration of study treatment), anytime between 0 to 15 minutes, 6 hours post-PCI and 24 hours post-PCI/discharge
Population: Safety Set included all participants in the FAS who received any study treatment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoints. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Micrograms per liter
  0 to 15 minutes Post-PCI: number analyzed (Participants) | 10 | 8 | 8
  0 to 15 minutes Post-PCI | -0.18 (0.290) | -0.18 (0.225) | -0.26 (0.490)
  6 Hours Post-PCI: number analyzed (Participants) | 9 | 8 | 6
  6 Hours Post-PCI | 0.70 (1.260) | 0.79 (2.208) | -0.63 (1.359)
  24 Hours Post- PCI/Discharge: number analyzed (Participants) | 6 | 1 | 3
  24 Hours Post- PCI/Discharge | -0.05 (0.804) | 31.80 (NA) — Standard deviation could not be calculated for only one participant. | 0.97 (0.643)

9. Secondary Outcome: Change From Baseline to Post-PCI for Cardiac Troponin I
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Microgram per liter
  0 to 15 minutes Post-PCI: number analyzed (Participants) | 10 | 8 | 8
  0 to 15 minutes Post-PCI | -0.04 (0.126) | 0.01 (0.035) | 0.04 (0.052)
  6 Hours Post-PCI: number analyzed (Participants) | 9 | 8 | 6
  6 Hours Post-PCI | 0.58 (1.310) | 0.13 (0.354) | 0.08 (0.204)
  24 Hours Post- PCI/Discharge: number analyzed (Participants) | 6 | 1 | 3
  24 Hours Post- PCI/Discharge | -0.03 (0.197) | 5.50 (NA) — Standard deviation could not be calculated for only one participant. | 0.30 (0.300)

10. Secondary Outcome: Number of Participants With Procedural Myocardial Injury
Description: Procedural myocardial injury was defined as elevation of cardiac troponin (cTn) values greater than (>) 99th percentile upper reference limit (URL) in participants with normal baseline values (<= 99th percentile URL) or elevation of cTn by > 20% of the baseline value in participants with elevated cTn levels (>99th percentile URL).
Time Frame: At 6 hours and 24 hours post-PCI/discharge on Day 1
Population: Safety Set included all participants in the FAS who received any study treatment. Combined data for Stage A and Stage B is presented as pre-specified in protocol. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here 'Number Analyzed' indicates number of participants evaluable at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  6 Hours Post-PCI: number analyzed (Participants) | 9 | 8 | 6
  6 Hours Post-PCI | 3 | 1 | 1
  24 Hours Post-PCI/Discharge: number analyzed (Participants) | 6 | 1 | 3
  24 Hours Post-PCI/Discharge | 1 | 1 | 2

11. Secondary Outcome: Concentration of Temanogrel
Description: Observed plasma concentration of temanogrel. Lower limit of quantification (LLOQ) of temanogrel was 0.500 nanograms/milliliter (ng/mL).
Time Frame: Pre-PCI, anytime between 0 to 15 minutes,1 hour, 3 hours, 6 hours post-PCI and 24 hours post PCI/discharge
Population: Pharmacokinetic (PK) set included all participants in the Safety Set with at least 1 post dose PK measurement. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoints. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg
Number analyzed (Participants) | 10 | 8
Nanograms per milliliter
  Pre-PCI: number analyzed (Participants) | 9 | 7
  Pre-PCI | 1558.3889 (2156.89423) | 1869.8571 (1815.65878)
  0 to 15 minutes post PCI: number analyzed (Participants) | 10 | 6
  0 to 15 minutes post PCI | 126.9900 (31.08320) | 265.0000 (109.83260)
  1 hour post PCI: number analyzed (Participants) | 6 | 6
  1 hour post PCI | 84.8667 (24.45278) | 134.1667 (36.56455)
  3 hours post PCI: number analyzed (Participants) | 6 | 7
  3 hours post PCI | 41.8500 (17.23969) | 87.1714 (90.12348)
  6 hours post PCI: number analyzed (Participants) | 9 | 8
  6 hours post PCI | 24.6522 (19.78224) | 36.9000 (14.94380)
  24 hours post-procedure/discharge: number analyzed (Participants) | 4 | 0
  24 hours post-procedure/discharge | NA (NA) — Data were not calculated as all values were below the limit of detection. |

12. Secondary Outcome: Concentration of AR295980
Description: Observed plasma concentration of AR295980.
Time Frame: Pre-PCI, anytime between 0 to 15 minutes,1 hour, 3 hours, 6 hours post-PCI and 24 hours post PCI/discharge
Population: PK set will include all participants in the Safety Set with at least 1 post dose PK measurement. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoints. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg
Number analyzed (Participants) | 10 | 8
Nanograms per milliliter
  Pre-PCI: number analyzed (Participants) | 9 | 7
  Pre-PCI | 1.0472 (0.87240) | 3.2010 (3.97562)
  0 to 15 minutes post PCI: number analyzed (Participants) | 10 | 6
  0 to 15 minutes post PCI | 6.3680 (2.61560) | 6.8183 (2.24211)
  1 hour post PCI: number analyzed (Participants) | 6 | 6
  1 hour post PCI | 5.0750 (1.81783) | 8.0783 (4.32397)
  3 hours post PCI: number analyzed (Participants) | 6 | 7
  3 hours post PCI | 3.6933 (1.18230) | 5.5300 (2.48489)
  6 hours post PCI: number analyzed (Participants) | 9 | 8
  6 hours post PCI | 2.4678 (0.79325) | 5.2650 (3.21979)
  24 hours post-PCI/discharge: number analyzed (Participants) | 4 | 0
  24 hours post-PCI/discharge | 0.3518 (0.40765) |

13. Secondary Outcome: Concentration of AR295981
Description: Observed plasma concentration of AR295981.
Time Frame: Pre-PCI, anytime between 0 to 15 minutes,1 hour, 3 hours, 6 hours post-PCI and 24 hours post PCI/discharge
Population: PK set included all participants in the Safety Set with at least 1 post dose PK measurement. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoints. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg
Number analyzed (Participants) | 10 | 8
Nanograms per milliliter
  Pre-PCI: number analyzed (Participants) | 9 | 7
  Pre-PCI | 1.8042 (1.11941) | 5.9129 (8.69909)
  0 to 15 minutes post PCI: number analyzed (Participants) | 9 | 6
  0 to 15 minutes post PCI | 0.9032 (0.46521) | 1.9030 (1.05032)
  1 hour post PCI: number analyzed (Participants) | 6 | 6
  1 hour post PCI | 0.6743 (0.36798) | 1.6575 (0.73395)
  3 hours post PCI: number analyzed (Participants) | 6 | 7
  3 hours post PCI | 0.4677 (0.37748) | 1.0651 (0.32193)
  6 hours post PCI: number analyzed (Participants) | 9 | 8
  6 hours post PCI | 0.2899 (0.35198) | 0.8685 (0.51239)
  24 hours post-PCI/discharge: number analyzed (Participants) | 4 | 0
  24 hours post-PCI/discharge | NA (NA) — Data were not calculated as all values were below the limit of detection. |

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: An adverse event (AE) was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start emerges. AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 as grade 1: mild; grade 2: moderate; grade 3: severe, grade 4: life threatening, grade 5: death related to AE. Number of participants with any TEAE and grade 3 or higher TEAE have been reported.
Time Frame: From start of study treatment on day 1 to up to maximum of 10 days
Population: The safety set included all participants in the FAS who received any study treatment. Combined data for Stage A and Stage B is presented as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  Any TEAE | 4 | 7 | 4
  Grade 3 or higher TEAE | 0 | 2 | 1

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events Leading to Discontinuation of Study Treatment and Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start emerges. SAE was an AE resulting in any of the following outcomes or considered medically significant: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or birth defect. Relatedness was based on investigator's assessment.
Time Frame: From start of study treatment on day 1 to up to maximum of 10 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  SAEs | 0 | 2 | 1
  Adverse events leading to discontinuation of study treatment | 0 | 0 | 0
  Treatment-Related TEAEs | 1 | 1 | 0

16. Secondary Outcome: Number of Participants With Treatment-Related TEAEs According to the Preferred Term
Description: An adverse event was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start emerges. Relatedness was based on investigator's assessment.
Time Frame: From start of study treatment on day 1 to up to maximum of 10 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 9
Participants
  Vascular access site haematoma | 1 | 0 | 0
  Hypertension | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment on Day 1 to up to maximum of 10 days
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other, or a participant may have experienced both serious and non-serious event.
Arm/Group | Temanogrel 20 mg | Temanogrel 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/8 | 1/9
Other Adverse Events (participants affected / at risk) | 4/10 | 7/8 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temanogrel 20 mg (N=10) | Temanogrel 40 mg (N=8) | Placebo (N=9)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temanogrel 20 mg (N=10) | Temanogrel 40 mg (N=8) | Placebo (N=9)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 4 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to a business decision that was not due to any safety concerns. The number of participants was smaller than originally planned and only summary statistics were therefore generated for primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT04848220/Prot_SAP_000.pdf